CLINICAL TRIAL: NCT05937867
Title: A Randomized, Double-blinded, Placebo-controlled，Phase II Clinical Study to Evaluate the Efficacy and Safety of HS-10353 in Participants With Postpartum Depression
Brief Title: A Phase II Study of HS-10353 in Participants With Postpartum Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10353-202
Record Dates: First submitted 2023-07-02; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10353 Capsules (Experimental)
  Interventions: Drug: HS-10353 Capsules 30 mg, Oral, QN for 14 days; Drug: HS-10353 Capsules 50 mg, Oral, QN for 14 days
- Placebo for HS-10353 Capsules (Experimental)
  Interventions: Drug: HS-10353 Capsules matching placebo, 30mg, Oral, QN for 14 days.; Drug: HS-10353 Capsules matching placebo, 50mg, Oral, QN for 14 days

INTERVENTIONS:
Drug: HS-10353 Capsules 30 mg, Oral, QN for 14 days — HS-10353 Capsules 30 mg
  Arms: HS-10353 Capsules
Drug: HS-10353 Capsules 50 mg, Oral, QN for 14 days — HS-10353 Capsules 50 mg
  Arms: HS-10353 Capsules
Drug: HS-10353 Capsules matching placebo, 30mg, Oral, QN for 14 days. — Placebo
  Arms: Placebo for HS-10353 Capsules
Drug: HS-10353 Capsules matching placebo, 50mg, Oral, QN for 14 days — Placebo
  Arms: Placebo for HS-10353 Capsules

SUMMARY:
The primary purpose of this study is to determine if treatment with HS-10353 reduces depressive symptoms in participants with postpartum depression (PPD) compared to placebo as assessed by the change from baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) total score at Day 15. And the secondary purpose of this study is to evaluate the safety and tolerability of HS-10353 compared to placebo as assessed by the incidence of adverse events, clinical laboratory evaluations, electrocardiogram (ECG) parameters, the Columbia Suicide Severity Rating Scale (C-SSRS), and the 20-item Physician Withdrawal Checklist (PWC-20).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18 to 45 years (including cut-off)
* Based on the investigator's clinical evaluation, subjects met the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) criteria for recurrent depressive disorder (MDD) or single episode MDD without psychotic symptoms, and the onset of this depression occurred between 28 weeks of gestation and 4 weeks postpartum
* ≤12 months post partum
* Hamilton Depression Scale (HAM-D17) total score ≥26
* Subjects who are not taking antidepressants for a current episode, or who have taken an oral antidepressant (SSRIs or SNRIs limited, including citalopram, Escitalopram, paroxetine, sertraline, venlafaxine, norvenlafaxine, duloxetine, Minapram) for at least 30 days at a pre-screening stable dose (allowing for a reduction of the drug within 1 week prior to screening),Or who had used any antidepressant before screening but had stopped taking it for at least five drug half-lives
* Agree to discontinue the use of other new antidepressants, antipsychotics, mood stabilizers, and benzodiazepine sedatives and hypnotics during administration
* According to the investigators, the subjects were generally in good physical condition, and no clinically significant abnormalities were found in physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, etc.) during screening
* Urine beta-human chorionic gonadotropin (beta-hCG) negative
* Agree to abstain from sex or other effective contraceptive methods for 30 days from screening until the last dose, and no egg donation plan is planned during this period
* If you have stopped breastfeeding, you must agree to stop breastfeeding before the first dose, and at least 7 days after the last dose.Able to communicate well with researchers, willing and able to comply with the lifestyle restrictions specified in the protocol, and cooperate with the completion of the experiment
* Subjects should fully understand the study content and process, as well as possible adverse reactions, and voluntarily sign an informed consent form (ICF).

Exclusion Criteria:

* Accompanied by psychotic symptoms
* In addition to depression, current history and previous history met the diagnostic criteria for other psychiatric disorders in the DSM-5 and were judged by the investigators to have potential implications for clinical studies
* Meet the diagnostic criteria for treatment-resistant depressive disorder
* Homicidal ideation/intent was present, or based on the Columbia Suicide Severity Assessment Scale (C-SSRS), the subject had a history of suicidal intent/self-harm behavior during the current depressive episode
* Atypical antipsychotics, mood stabilizers (e.g., olanzapine, risperidone, quetiapine, aripiprazole, iprazole, Ziprasidone, calilrazine, sodium valproate, lithium carbonate) were used during the current depressive episode.
* History of modified electrical tics (MECT), transcranial magnetic stimulation (TMS), or prior treatment with vagus nerve stimulation (VNS) or deep brain stimulation (DBS) within 1 month prior to screening
* Present or previous history of disease or dysfunction affecting clinical trials, including but not limited to nervous system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal musculoskeletal system, metabolic endocrine system, skin disease, blood system disease, immune disease and tumor, clinically significant chronic disease or poor disease control,The researchers assessed that they were not fit to participate in this study
* The presence of any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or that may pose a hazard to the subjects participating in the trial;Such as gastrointestinal surgery history (gastrectomy, gastrostomy, enterectomy, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcer, gastrointestinal bleeding history, etc
* Previous history of seizures (except convulsions caused by febrile convulsions in children)
* History of severe allergies
* A history of drug abuse or benzodiazepine dependence within the last 1 year
* A history of alcohol abuse in the last 6 months (i.e. drinking more than 14 standard units per week, 1 unit =360ml beer or 45ml spirits with 40% alcohol or 150ml wine)
* Participate in any clinical study within 30 days prior to screening
* Take CYP3A4, CYP2C9, or CYP2C19 suppressants (e.g. Clarithromycin, itraconazole, ketoconazole, voriconazole, fluvoxamine, fluconazole, fluoxetine, ticlopidine) for 14 days prior to first dosing (or 5 half-lives, whichever is longer) and throughout the study period.Or grapefruit/grapefruit juice, grapefruit/grapefruit, Seville orange or products rich in such substances
* CYP inducers such as rifampin, carbmazepine, Ritonavir, enzalutamide, efavirenan, nevirapine, phenytoin, phenobarbital, or St. John's Wort were taken within 14 days prior to first administration (or 5 half-lives, whichever is longer) and throughout the study period
* 12-lead electrocardiogram and other test indicators abnormal and clinically significant, such as: Friericia corrected QT interval (QTcF= QT/RR0.33), absolute value > 470ms
* Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), syphilis seroresponse (TRUST) positive
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN), serum creatinine (Cr) > 1.5 times ULN
* Poor compliance or other problems, the researcher considered it inappropriate to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the HAM-D17 total score at day 15 | Baseline, Day 15
  The HAM-D17 is used to rate the severity of depression in participants who are already diagnosed as depressed. The HAM-D17 total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. Higher scores indicated more severe depression. A negative change from baseline indicates less depression

SECONDARY OUTCOMES:
Change From Baseline in the HAM-D Total Score at Days 3, 8, 21 and 28 | Baseline, Day 3, Day 8, Day 21, Day 28
  The HAM-D17 is used to rate the severity of depression in participants who are already diagnosed as depressed. The HAM-D17 total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. Higher scores indicated more severe depression. A negative change from baseline indicates less depression
Percentage of Participants With HAM-D17 Response | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  HAM-D17 Response was defined as having a 50 percent (%) or greater reduction from Baseline in HAM-D17 total score. The HAM-D17 total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. Higher scores indicated more depression.
Percentage of Participants With HAM-D17 Remission | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  HAM-D17 Remission was defined as a HAM-D17 total score of less than or equal to (<=)7. The HAM-D17 total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52.
Change From Baseline in the Clinical Global Impressions - Severity Scale (CGI-S) Total Score | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  The CGI-S is a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis. A participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7= extremely ill participants. A lower score indicates a better outcome. A negative change from baseline indicates improvement. MMRM was used for the analysis
Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  The Clinical Global Impression - Improvement (CGI-I) item of the CGI scale uses a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. CGI response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved). The percentage of participants with overall improvement in post-treatment condition, rated by investigator as very much improved (CGI-I score of 1) or much improved (CGI-I score of 2) is reported.
Change From Baseline in Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  The MADRS is a 10-item questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item was scored in a range of 0 (no symptoms) to 6 (symptoms of maximum severity). The MADRS total score was calculated as the sum of the 10 individual item scores and could range from 0 to 60. Higher scores indicated more severe depression. A negative change from Baseline indicates less depression.
Change From Baseline in Self-Reported Measures of Depressive Symptoms, as Assessed by the Edinburgh Postnatal Depression Scale (EPDS) Total Score | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  The EPDS is a self-rated depressive symptom severity scale specific to the perinatal period which consists of 10 individual items. Each item is rated on a 4-point scale ranging from 0 to 3 points. The EPDS total score is calculated as the sum of the 10 individual item scores, ranging from 0 points to 30 points with a higher score indicating more depression. A negative change indicates improvement.
Change From Baseline in Self-Reported Measures of Depressive Symptoms, as Assessed by the 9-item Patient Health Questionnaire (PHQ-9) Score | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  The PHQ-9 is a self-rated depressive symptom severity scale to monitor severity over time for newly diagnosed participants or participants in current treatment for depression. Scoring was based on participants responses to 9 specific questions as follows: 0 = not at all; 1 = several days; 2 = more than half the days; and 3 = nearly every day. The score were calculated as the sum of the 9 individual item scores. The PHQ-9 total score was categorized as follows: 1 to 4 = minimal depression, 5 to 9 = mild depression, 10 to 14 = moderate depression, 15 to 19 = moderately severe depression; and 20 to 27 = severe depression. The PHQ-9 total score ranges from 1 to 27 with a higher score indicating more depression. A negative change from baseline indicates reduced depression. MMRM was used for the analysis.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score | Baseline, Day 3, Day 8, Day 15, Day 21, Day 28
  The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The individual items were scored in a range of 0 (not present) to 4 (very severe). The HAM-A total score was calculated as the sum of the 14 individual item scores and could range from 0 to 56 where a score of <17=mild severity; 18-24= mild to moderate severity and 25-30=moderate to severe severity. A negative change from Baseline indicates less anxiety.
Change From Baseline in (PWC-20) Total Score | Baseline, Day 15, Day 21
Number of Participants With adverse events (AEs), serious adverse events (SAEs), and adverse events leading to withdrawal from the trial, and association with the investigational drug | Up to Day 28
  An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE with an onset that occurs after receiving study drug.
Number of Participants With Potentially Clinically Significant Vital Sign Measurements | Up to Day 28
  Vital signs included assessments of systolic blood pressure (SBP), diastolic blood pressure (DBP), temperature, respiration and heart rate.
Number of Participants With Potentially Clinically Significant Laboratory Evaluations | Up to Day 28
  ECG parameters included assessment of the standard 12-lead ECG intervals: QT, QTcF, PR, RR, QRS, and heart rate. Heart rate was measured in terms of beats per minute. Change from Baseline in heart rate, PR Interval, RR Interval, QRS Duration, QT Interval, QTcF Interval is reported.

IPD SHARING:
Plan to Share IPD: No